CLINICAL TRIAL: NCT07123116
Title: Shenbai Granules for Preventing Recurrence of Low-Risk Colorectal Adenomas: A Multicenter Randomized Controlled Clinical Trial
Brief Title: Shenbai Granules for Preventing Recurrence of Low-Risk Colorectal Adenomas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The Second Hospital of Shandong University (Other); Shengjing Hospital (Other); Shenzhen Hospital of Southern Medical University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Sichuan Provincial People's Hospital (Other); Shanxi Provincial People's Hospital (Other Government); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025NL-108-02
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Adenoma; TCM; Low Risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shenbai Granules (Experimental): Shenbai Granules is a traditional Chinese medicine preparation formulated from eight herbal ingredients, including Sophorae Flavescentis Radix (Kushen), Coptidis Rhizoma (Huanglian), and other herbs. It exerts therapeutic effects by clearing heat and drying dampness, while simultaneously invigorating the spleen and replenishing qi.
  Interventions: Drug: Shenbai Granules
- Placebo (Placebo Comparator): The placebo was formulated using Shenbai Granules dry extract powder at 2% (w/w) of the equivalent dose found in the compound herbal granules, supplemented with colorants and flavoring agents to ensure visual and gustatory consistency with the Shenbai Granules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Shenbai Granules — Dosage: bag 10g per , administered twice daily continuously for 180 days.
  Arms: Shenbai Granules
Drug: Placebo — Dosage: 10g per bag, administered twice daily continuously for 180 days.
  Arms: Placebo

SUMMARY:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Shenbai Granules for Preventing Recurrence of Low-Risk Colorectal Adenomas（LRCRA）.

Study Population: Post-resection patients with low-risk colorectal adenomas and Spleen Deficiency with Dampness-Heat Syndrome per TCM criteria.

Sample Size: 450 subjects (1:1 randomization; 225 per arm) accounting for ≤20% dropout.

Study Hypothesis (Exploratory) ： This exploratory trial aims to evaluate the potential efficacy and safety of Shenbai Granules, a TCM formula, in reducing LRCRA recurrence. Based on preliminary data suggesting a 32.64% relative risk reduction in LRCRA recurrence at 2 years, we hypothesize that Shenbai Granules may demonstrate clinically meaningful prevention of adenoma recurrence and offer a favorable safety profile in the target TCM syndrome population. No formal statistical hypothesis is tested.

Statistical Analysis Analysis Sets: mITT (primary efficacy), PPS, SS (safety). Primary Analysis: Proportion difference (Newcombe method) and χ²/Fisher's exact test (stratified CMH if applicable).

Sensitivity analyses: PPS, tipping-point imputation for missing data. Safety: Descriptive summaries of AEs/SAEs (MedDRA-coded), lab abnormalities.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, all of the following inclusion criteria must be met:

1. Aged 40-75 years, regardless of sex;
2. Patients with histologically confirmed high-risk adenomas undergoing initial polypectomy, with high-quality colonoscopy performed within 14 days before randomization;
3. Complete resection of all detected lesions during colonoscopy;
4. Meeting TCM diagnostic criteria for spleen deficiency with dampness-heat syndrome;
5. Provision of signed informed consent and ability to comply with long-term follow-up.

   1. High-quality colonoscopy is defined as: Boston Bowel Preparation Scale (BBPS) score ≥6, cecal intubation with photo-documentation and withdrawal time ≥6 minutes. If quality standards cannot be confirmed, a repeat colonoscopy is required.

      -

      Exclusion Criteria:

      Subjects who meet any of the following exclusion criteria will not be enrolled in this study:

1) Complicated with malignant tumor or having a history of malignant tumor; 2) Personal or family history of familial polyposis or hereditary nonpolyposis colorectal cancer; 3) History of inflammatory bowel disease; 4) Suffering from malignant tumors of other systems except the study disease within 5 years before screening, except for malignant tumors that have been cured after treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery); 5) Complicated with severe organic diseases such as cardiovascular and cerebrovascular diseases, autoimmune diseases, diseases of the motor, hematological, digestive, respiratory, immune, circulatory, reproductive, urinary, or endocrine systems, or patients with neuropsychiatric diseases, abnormal coagulation function, severe postoperative complications, such as gastrointestinal bleeding, perforation, cholangitis, abdominal infection, cardiopulmonary function depression, mesenteric laceration, or pneumoperitoneum, etc., or other acute and chronic diseases that may affect treatment and prognosis; those with Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) levels exceeding 2.5 times the upper limit of normal, Alkaline Phosphatase (ALP) levels exceeding 2 times the upper limit of normal, or abnormal electrocardiogram results assessed by investigators as clinically significant; 6) Patients with active gastrointestinal diseases, at risk of gastrointestinal perforation, or suffering from other diseases that can significantly interfere with the absorption, distribution, metabolism, or excretion of the trial drug, such as inability to take oral drugs, uncontrolled nausea or vomiting, intestinal obstruction, chronic diarrhea due to extensive intestinal resection, Crohn's disease, ulcerative colitis, or chronic diarrhea, etc.; 7) Having used the following treatments that may have a preventive effect on colorectal adenomas within 3 months before screening, for 3 consecutive months, at least 2 times a week, with an interruption time of less than 2 weeks: taking non-steroidal anti-inflammatory drugs such as aspirin, ibuprofen, celecoxib, etc, metformin, berberine hydrochloride, folic acid, vitamin D, selenium supplements, and calcium supplements, or maintaining systemic immunotherapy, or using Chinese patent medicines based on the indications in the instructions or Chinese herbal decoctions with the effects of invigorating spleen and replenishing qi, clearing heat and eliminating dampness; those who have undergone a washout period of 1 month or 5 half-lives of the drug whichever is longer can be enrolled; 8) Those with cold syndrome such as fear of cold, cold pain in the waist and abdomen, cold limbs, and preference for hot drinks when thirsty; 9) Pregnant or lactating women, as well as men or women of childbearing age who have plans for childbearing recently or within 7 months before the study; 10) Having participated in, or currently participating in, other clinical trials of drugs or research devices within 1 month before screening or within 5 half-lives of the trial drug whichever is longer, or planning to participate in any other clinical trials during this study; 11) Allergic constitution with a history of allergy to two or more drugs or foods or known allergy to the components of the study drug; 12) Other conditions deemed unsuitable for inclusion by the investigator, such as expected poor compliance, cognitive impairment, etc.

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Detection rate of metachronous colorectal adenoma within 3 years after initial administration. | 3 years
  the proportion of patients with detected metachronous colorectal adenomas during surveillance colonoscopy performed within 3 years after baseline polypectomy or adenoma resection to the total number of patients in the group.

SECONDARY OUTCOMES:
Cumulative number, quantity, size, location, and pathology of detected metachronous colorectal adenomas within 3 years after initial administration. | 3 years
  The cumulative number, mean number, mean size, location distribution (left-sided colon, right-sided colon, rectum), and histological classification (histological architecture: tubular adenoma, villous adenoma, tubulovillous adenoma; dysplasia grade: high-grade intraepithelial neoplasia [HGIN], low-grade intraepithelial neoplasia [LGIN]) of metachronous colorectal adenomas detected during surveillance colonoscopy performed within 3 years after baseline polypectomy.
Detection rate of serrated lesions within 3 years after initial administration. | 3 years
  The proportion of patients with detected serrated lesions during surveillance colonoscopy performed within 3 years after baseline polypectomy or adenoma resection to the total number of patients in the group.
Cumulative number, quantity, size, location, and pathology of detected serrated lesions within 3 years after initial administration. | 3 years
  The cumulative number, mean number, mean size, location distribution (left-sided colon, right-sided colon, rectum), and histological classification (Traditional Serrated Adenoma [TSA], Sessile Serrated Lesion [SSL], Hyperplastic Polyp [HP]) of serrated lesions detected during surveillance colonoscopy performed within 3 years after baseline polypectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China